CLINICAL TRIAL: NCT01772862
Title: Rehabilitation Including Social and Education in Children and Teenagers With Cancer
Brief Title: Rehabilitation Including Social and Physical Activity in Children and Teenagers With Cancer
Acronym: RESPECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kjeld Schmiegelow (Other)
Collaborators: Odense University Hospital (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Kjeld Schmiegelow, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RESPECT - physical activity; H-3-2012-105 (Other: Ethical Review Board of Region Hovedstaden)
Record Dates: First submitted 2013-01-11; First posted 2013-01-21 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Childhood Cancer
Keywords: childhood; cancer; physical activity; quality of life
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Only conventional supportive care (No Intervention): The children receive conventional supportive care with respect to physical training
- Intervention group (Experimental): The intervention components includes (real time sequence):
  An educational session where the child is educated on his/her cancer disease. An education session in the child's school where the child´s teachers, classmates and their parents are educated on the child´s cancer disease.
  Appointment of two classmates as "ambassadors". An individualized physical training program combining supervised and non-supervised training 3-5 times per week.
  Continued specialized physical training when relevant. At two weeks intervals joined education, physical and social activity days at the hospital with together with one of the ambassadors
  Interventions: Behavioral: Intervention group

INTERVENTIONS:
Behavioral: Intervention group — The intervention components includes (real time sequence):
  An educational session where the child is educated on his/her cancer disease. An education session in the child's school where the child´s teachers, classmates and their parents are educated on the child´s cancer disease.
  Appointment of two classmates as "ambassadors". An individualized physical training program combining supervised and non-supervised training 3-5 times per week.
  Continued specialized physical training when relevant. At two weeks intervals joined education, physical and social activity days at the hospital with together with one of the ambassadors
  Other Names: Integrated physical training
  Arms: Intervention group

SUMMARY:
The purpose of this study is to determine whether early rehabilitation intervention including individualized physical training and social activities with a class mate at two weeks intervals at the ped.onc. center will increase children with cancer's level of physical performance

DETAILED DESCRIPTION:
Background In Denmark 200 children under the age of 18 are diagnosed annually with cancer and the prevalence of patients undergoing anticancer therapy is 300. The expected five-year survival rate is 80%, but since the treatment is intensive with a high risk of life-threatening infections, these patients are frequently isolated at home or in hospital during their 1-2 years of therapy, which means reduced contact with their normal school environment, leisure activities and friends. Long-term survivors of childhood cancer frequently have compromised age-appropriate social relationships and psychosocial development, difficulties with resuming physical activities, and poor self-esteem leading to reduced quality of life. Intervention studies designed to improve physical and social function during treatment of children with cancer are lacking.

Aim To develop an interactive rehabilitation programme that a) preserve the educational, physical and psychosocial life of the patients or even obtains "growth with cancer", b) maintains the child's everyday life (e.g. normal social relationships), and c) improves long-term physical performance, social competences, higher grade educational enrollment, and later integration into the labour market.

Theoretical basis This project is inspired by Erving Goffman's interactional theory on normality and related concepts of stigma and frame analysis as well as Thomas Scheff's theory on the concept of emotional and social bonds and the development of the sociology of emotions.

Material and methods Intervention group: Children aged 6.0-18.0 years diagnosed with cancer 2013-2015 at Rigshospitalet (covers eastern part of Denmark (approximately 50% of total population)).

Control group:

The primary control group is children with cancer treated at the university hospitals in Odense, Aarhus and Aalborg 2013-2015.

In addition, outcome data for cases will be compared with three other (secondary) comparative groups: a) children with cancer treated at any Danish childhood oncology unit throughout Denmark in 2012 (historical controls); b) the sibling closest in age to the intervention group patients (family matched); and c) the intervention group patient's classmates.

Physical performance end point The physical performance will be monitored by: Andersen interval test, Timed up and go test, Sit to stand test, flamingo balance test, strength of hand by squeeze dynamometer and VO2 peak sub-max test.

Physical measures

Dexa scan

Questionnaires: PedsQL, Strength and Difficulties Questionnaire (SDQ), Revised Child anxiety and Depression Scale, Resilience, Loneliness and Social Dissatisfaction Questionnaire og The Children´s Impact of Event Scale 13.

Qualitative interviews: Qualitative interviews are performed with children with cancer, their parents, and the ambassadors. The focus will be on sociometric status, social independence and competences, self-esteem, fatigue, physical activity, educational outcome, and safety issues as well as an evaluation of the intervention program.

Outcomes and statistical considerations Provided all children with cancer (6-18 years) are included in the intervention or control group this study will be national cohort study including approximately 120 intervention children and 120 control children during the three year intervention period.

In relation to physical performance the power calculation is based on previous published small studies that found a baseline VO2peak of 24.3 (SD5.9) among children with ALL. If 120 children are included in the intervention and in the control group, then it the study will have a power or more than 0.85 to detect a 10% improvement and a power of 0.95 to detect a 15% improvement.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with cancer and treated at the pediatric oncology units in Denmark (Rigshospitalet, Odense University hospital, Aarhus University Hospital and Aalborg University Hospital)

Children diagnosed with non-malignant diseases treated with surgery, chemotherapy or irradiation similar to cancer (e.g. benign CNS tumors, langerhans cell histiocytosis, Myelodysplastic Syndrome (MDS)) and treated at the pediatric oncology units in Denmark (Rigshospitalet, Odense University hospital, Aarhus University hospital and Aalborg University Hospital).

Attend school at the time of diagnosis

Able to communicate in Danish

Exclusion Criteria:

* Mental retardation at the time of diagnosis (including Down syndrome) Terminal illness at the time of diagnoses Severe co-morbidity

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Level of VO2 max | 1 year after cessation of first-line cancer treatment
  We hypothesize that the children in the intervention group receiving a individualized physical training program three time a week during the intensive treatment period with surgery, irradiation or chemotherapy treatments will have a 10% higher VO2max level than children with cancer in the control group who do not receive such training

SECONDARY OUTCOMES:
Health quality of life | Diagnosis, 6 months after diagnoses, 1 year post treatment
  Quality of life is assessed by questionnaires, and qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Schmiegelow, M.D, Study Director — University Hospital of Copenhagen, Rigshospitalet
Locations (1):
- Kjeld Schmiegelow, Copenhagen, Denmark

REFERENCES:
- [Derived] Nielsen MKF, Christensen JF, Frandsen TL, Thorsteinsson T, Andersen LB, Christensen KB, Wehner PS, Hasle H, Adamsen LO, Schmiegelow K, Larsen HB. Effects of a physical activity program from diagnosis on cardiorespiratory fitness in children with cancer: a national non-randomized controlled trial. BMC Med. 2020 Jul 6;18(1):175. doi: 10.1186/s12916-020-01634-6. PMID 32624004
- [Derived] Nielsen MKF, Christensen JF, Frandsen TL, Thorsteinsson T, Andersen LB, Christensen KB, Nersting J, Faber M, Schmiegelow K, Larsen HB. Testing physical function in children undergoing intense cancer treatment-a RESPECT feasibility study. Pediatr Blood Cancer. 2018 Aug;65(8):e27100. doi: 10.1002/pbc.27100. Epub 2018 May 9. PMID 29741279
- [Derived] Thorsteinsson T, Larsen HB, Schmiegelow K, Thing LF, Krustrup P, Pedersen MT, Christensen KB, Mogensen PR, Helms AS, Andersen LB. Cardiorespiratory fitness and physical function in children with cancer from diagnosis throughout treatment. BMJ Open Sport Exerc Med. 2017 May 12;3(1):e000179. doi: 10.1136/bmjsem-2016-000179. eCollection 2017. PMID 28761697
- [Derived] Lindgren LH, Schmiegelow K, Helms AS, Thorsteinsson T, Larsen HB. In sickness and in health: classmates are highly motivated to provide in-hospital support during childhood cancer therapy. Psychooncology. 2017 Jan;26(1):37-43. doi: 10.1002/pon.4094. Epub 2016 Feb 12. PMID 26872002
- [Derived] Thorsteinsson T, Helms AS, Adamsen L, Andersen LB, Andersen KV, Christensen KB, Hasle H, Heilmann C, Hejgaard N, Johansen C, Madsen M, Madsen SA, Simovska V, Strange B, Thing LF, Wehner PS, Schmiegelow K, Larsen HB. Study protocol: Rehabilitation including Social and Physical activity and Education in Children and Teenagers with Cancer (RESPECT). BMC Cancer. 2013 Nov 14;13:544. doi: 10.1186/1471-2407-13-544. PMID 24229362